CLINICAL TRIAL: NCT04316728
Title: Clinical Performance of the VivaDiag ™ COVID-19 lgM / IgG Rapid Test in a Cohort of Negative Patients for Coronavirus Infection for the Early Detection of Positive Antibodies for COVID-19
Brief Title: Clinical Performance of the VivaDiag ™ COVID-19 lgM / IgG Rapid Test in Early Detecting the Infection of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Studi Internazionali, Italy (Network)
Collaborators: VivaChek Laboratories, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VivaDiag-2020
Record Dates: First submitted 2020-03-14; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Infections
Keywords: COVID-19; IgM Test; IgG Test
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- negative Patients (Other): Adult HCWs with no signs or symptom of coronavirus infection and no known previous history of contact with patients positive for COVID-19, working in a primary care setting and Adult patients with at least 2 chronic medical conditions routinely attending a General Practioner (GP) practice or an outpatients departments or a primary care facility
  Interventions: Device: VivaDiag™ COVID-19 lgM/IgG Rapid Test

INTERVENTIONS:
Device: VivaDiag™ COVID-19 lgM/IgG Rapid Test — VivaDiag™ COVID-19 lgM/IgG Rapid Test is an in vitro diagnostic for the qualitative determination of COVID-19 IgM and IgG antibodies in human whole blood (from vein or fingertip), serum or plasma

SUMMARY:
This study aim to evaluate the immune response of negative patients during a COVID-19 outbreak.

Patients are serially tested with a VivaDiag ™ COVID-19 lgM / IgG Rapid Test to evaluate the immune response in negative patients and the reliability of the test in those patients who develop clinical signs of COVID-19 during the trial.

DETAILED DESCRIPTION:
This study aim to evaluate the immune response of negative patients during a COVID-19 outbreak in patients with no symptoms and with no known exposure to the COVID-19.

Patients are tested with a VivaDiag ™ COVID-19 lgM / IgG Rapid Test at day 0, day 7 and day 14. The investigators expect test to be negative on all the measurements in those patients that do not develop symptoms and that continue to have no known history of exposure to COVID-19

Patients that develop symptoms (cough, fever or respiratory distress) and a possible contact with people positive for COVID-19 OR patients that show a positive VivaDiag test during the time frame of the test are asked to attend the COVID-19 RT - PCR &CT.

Subsequently, the investigators will continue, repeating two tests seven days apart every 30 days (predefined times 0-7-14, then 30-37, 60-67) for the next six months. The investigators can evaluate to stop the test however before the six months if there are no new cases of COVID-19 for at least 21 days in the region where the enrolled patients live.

The test in use is the VivaDiag ™ COVID-19 lgM / IgG

Procedure (as per the protocol in use for the administration of the test)

1. take out the test kit and leave it at least 30 minutes in the room where the test will be performed.
2. place the test equipment on a clean and dust-free surface
3. First insert 10µL of whole blood or serum or plasma in the area reserved for blood (in the well) present on the test, then apply 2 drops of buffer.
4. read the result after 15 minutes

Interpretation of test results

Positive result

1. The anti-COVID-19 lgM antibody is detected if: the quality control band C and the lgM band are both colored and the lgG band does not stain. This means that the anti-COVID-19 lgM antibody is positive.
2. The anti-COVID-19 lgG antibody is detected if: the quality control band C and the lgG band are both colored and the lgM band does not stain. This means that the COVID-19 lgG antibody is positive.
3. The lgG and lgM anti-COVID-19 antibodies are detected if: the C band, the lgG band and the lgM band are all three colored. This means that the anti-COVID-19 lgG and lgM antibodies are both positive.

Negative result The anti-COVID-19 lgG and lgM antibodies are not detected if only the quality control C band is stained but the lgG and lgM bands are not colored, this means that the test is negative.

Invalid result

If the quality control band C does not color, regardless of whether the lgG and lgM bands are colored or not, the result is invalid and the test must be started again.

Specs of the test

Product Name VivaDiag™ COVID-19 IgM/IgG Rapid Test Test Principle Colloidal gold Sample Type Whole blood (from vein or fingertip), serum or plasma Sample Volume 10 μL Test Time 15 min Operation Temperature 18-25ºC Storage Temperature 2-30ºC Shelf Life (Unopened) 12 months

ELIGIBILITY:
Inclusion Criteria:

* Adults healthcare workers (HCW) OR
* Chronic patients with at least 2 chronic medical conditions

Exclusion Criteria:

* People that have been in contact with people positive for COVID-19 in the previous 14 days
* People with body temperature >37.5°C
* People with Dry cough
* People with Respiratory distress (Respiratory Rate >25/min or O2 Saturation <92%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with constant negative results | 30 days
  Number of patients with negative results in the three measurements, compared to the number of patients with at least one positive test
Number of patients with positive test with a positive PCR for COVID-19 | 30 days
  Number of patients that present at least one positive VivaDiag test that when subsequently tested with PCR remain positive
Overall Number of patients positive for COVID-19 | six months
  Where available, number of patients positive for COVID-19 IgG and IgM and positive for COVID-19 PCR
Overall Number of patients negative for COVID-19 | six months
  Where available, number of patients negative for COVID-19 IgG and IgM and negative for COVID-19 PCR
Number of patients with contrasting results | 30 days
  Where available, number of patients positive for COVID-19 IgG and IgM and negative for COVID-19 PCR, or negative for COVID-19 IgG and IgM and positive for COVID-19 PCR

SECONDARY OUTCOMES:
Reliability of the test | 30 days
  Number of Invalid results
Positive HCW | 60 days
  Number of healthcare workers that become positive for COVID-19 IgM or IgG
Number of Chronic Patients | 60 days
  Number of Chronic Patients that become positive for COVID-19 IgM or IgG

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Cipolla, MD, Study Director — Medical director of UCCP CATANZARO, Italy
Locations (1):
- Unità' Complesse di cure primarie (UCCP), ASP Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Still under development
Supporting Information: Study Protocol, CSR
Time Frame: 12 months
Access Criteria: Still under development

REFERENCES:
- [Background] Zarocostas J. What next for the coronavirus response? Lancet. 2020 Feb 8;395(10222):401. doi: 10.1016/S0140-6736(20)30292-0. No abstract available. PMID 32035538
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Phan LT, Nguyen TV, Luong QC, Nguyen TV, Nguyen HT, Le HQ, Nguyen TT, Cao TM, Pham QD. Importation and Human-to-Human Transmission of a Novel Coronavirus in Vietnam. N Engl J Med. 2020 Feb 27;382(9):872-874. doi: 10.1056/NEJMc2001272. Epub 2020 Jan 28. No abstract available. PMID 31991079
- [Background] Perlman S. Another Decade, Another Coronavirus. N Engl J Med. 2020 Feb 20;382(8):760-762. doi: 10.1056/NEJMe2001126. Epub 2020 Jan 24. No abstract available. PMID 31978944
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Gralinski LE, Menachery VD. Return of the Coronavirus: 2019-nCoV. Viruses. 2020 Jan 24;12(2):135. doi: 10.3390/v12020135. PMID 31991541
- [Background] Ronco C, Navalesi P, Vincent JL. Coronavirus epidemic: preparing for extracorporeal organ support in intensive care. Lancet Respir Med. 2020 Mar;8(3):240-241. doi: 10.1016/S2213-2600(20)30060-6. Epub 2020 Feb 6. No abstract available. PMID 32035509
- [Background] Lan L, Xu D, Ye G, Xia C, Wang S, Li Y, Xu H. Positive RT-PCR Test Results in Patients Recovered From COVID-19. JAMA. 2020 Apr 21;323(15):1502-1503. doi: 10.1001/jama.2020.2783. PMID 32105304
- [Background] Kobayashi T, Jung SM, Linton NM, Kinoshita R, Hayashi K, Miyama T, Anzai A, Yang Y, Yuan B, Akhmetzhanov AR, Suzuki A, Nishiura H. Communicating the Risk of Death from Novel Coronavirus Disease (COVID-19). J Clin Med. 2020 Feb 21;9(2):580. doi: 10.3390/jcm9020580. PMID 32098019
- [Background] Chan JF, Yip CC, To KK, Tang TH, Wong SC, Leung KH, Fung AY, Ng AC, Zou Z, Tsoi HW, Choi GK, Tam AR, Cheng VC, Chan KH, Tsang OT, Yuen KY. Improved Molecular Diagnosis of COVID-19 by the Novel, Highly Sensitive and Specific COVID-19-RdRp/Hel Real-Time Reverse Transcription-PCR Assay Validated In Vitro and with Clinical Specimens. J Clin Microbiol. 2020 Apr 23;58(5):e00310-20. doi: 10.1128/JCM.00310-20. Print 2020 Apr 23. PMID 32132196
- [Background] Zu ZY, Jiang MD, Xu PP, Chen W, Ni QQ, Lu GM, Zhang LJ. Coronavirus Disease 2019 (COVID-19): A Perspective from China. Radiology. 2020 Aug;296(2):E15-E25. doi: 10.1148/radiol.2020200490. Epub 2020 Feb 21. PMID 32083985
- [Background] Xiao Y, Torok ME. Taking the right measures to control COVID-19. Lancet Infect Dis. 2020 May;20(5):523-524. doi: 10.1016/S1473-3099(20)30152-3. Epub 2020 Mar 5. No abstract available. PMID 32145766
- [Background] Wang Y, Kang H, Liu X, Tong Z. Combination of RT-qPCR testing and clinical features for diagnosis of COVID-19 facilitates management of SARS-CoV-2 outbreak. J Med Virol. 2020 Jun;92(6):538-539. doi: 10.1002/jmv.25721. Epub 2020 Mar 11. No abstract available. PMID 32096564
- [Background] Li Y, Xia L. Coronavirus Disease 2019 (COVID-19): Role of Chest CT in Diagnosis and Management. AJR Am J Roentgenol. 2020 Jun;214(6):1280-1286. doi: 10.2214/AJR.20.22954. Epub 2020 Mar 4. PMID 32130038
- [Background] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Background] Zhang S, Diao M, Yu W, Pei L, Lin Z, Chen D. Estimation of the reproductive number of novel coronavirus (COVID-19) and the probable outbreak size on the Diamond Princess cruise ship: A data-driven analysis. Int J Infect Dis. 2020 Apr;93:201-204. doi: 10.1016/j.ijid.2020.02.033. Epub 2020 Feb 22. PMID 32097725
- [Background] Lippi G, Plebani M. Laboratory abnormalities in patients with COVID-2019 infection. Clin Chem Lab Med. 2020 Jun 25;58(7):1131-1134. doi: 10.1515/cclm-2020-0198. No abstract available. PMID 32119647
- [Background] Binnicker MJ. Emergence of a Novel Coronavirus Disease (COVID-19) and the Importance of Diagnostic Testing: Why Partnership between Clinical Laboratories, Public Health Agencies, and Industry Is Essential to Control the Outbreak. Clin Chem. 2020 May 1;66(5):664-666. doi: 10.1093/clinchem/hvaa071. No abstract available. PMID 32077933
- [Background] Habibi R, Burci GL, de Campos TC, Chirwa D, Cina M, Dagron S, Eccleston-Turner M, Forman L, Gostin LO, Meier BM, Negri S, Ooms G, Sekalala S, Taylor A, Yamin AE, Hoffman SJ. Do not violate the International Health Regulations during the COVID-19 outbreak. Lancet. 2020 Feb 29;395(10225):664-666. doi: 10.1016/S0140-6736(20)30373-1. Epub 2020 Feb 13. No abstract available. PMID 32061311